CLINICAL TRIAL: NCT02631057
Title: Comparison of the Length of Stay in Patients Hospitalized and Initiated With Dabigatran or Warfarin for a Concomitant Non-Valvular Atrial Fibrillation in Real-world Japanese Therapeutic Practice (SHORT-J)
Brief Title: Length of Stay in NVAF Patients Hospitalized and Initiated With Dabigatran or Warfarin in Japan
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.254
Record Dates: First submitted 2015-12-08; First posted 2015-12-15 (Estimated); Results first posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Non-Valvular Atrial Fibrillation
  Interventions: Drug: Dabigatran
- acute ischemic stroke
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Dabigatran — Dabigatran 110 mg capsule twice a day or 75 mg x 2 capsules twice a day
  Groups: Non-Valvular Atrial Fibrillation
Drug: Warfarin — Warfarin tablet (adjustment by each patients)
  Groups: acute ischemic stroke

SUMMARY:
The primary objective of this study is to compare the Length of Stay from treatment of oral anticoagulant initiation to hospital discharge of patients hospitalized and subsequently treated with dabigatran or warfarin for non-valvular atrial fibrillation in a real-world Japanese clinical practice. The secondary objective of the study is to compare LoS of patients hospitalized with 1) acute ischemic stroke, and 2) due to non-valvular atrial fibrillation. Other objectives are (1) to compare the in-hospital direct and indirect-related costs between dabigatran and warfarin, and (2) to compare the rates of patients directly discharged at home after the index hospitalization between dabigatran and warfarin.

ELIGIBILITY:
Inclusion criteria:

1. Hospitalized patients among patients having a visit record with a confirmed diagnosis of NVAF (ICD-10 Code: I48) and prescribed dabigatran or warfarin in the hospitalization period

Exclusion criteria:

1. Having a record with a diagnosis of atrial flutter, valvular atrial fibrillation or postoperative atrial fibrillation diagnosis as standard disease name during the study period.
2. Having a record with a diagnosis of rheumatic atrial fibrillation (ICD-10 code I05 to I09 [chronic rheumatic atrial fibrillation])or mechanical-valvular atrial fibrillation (ICD-10 code T820 [artificial cardiac valve mechanical complication]) during the study period.
3. Having a record with a confirmed diagnosis of cancer (ICD-10 code C00-C97 [malignant neoplasm]) during the study period.
4. Having a record of dialysis (class J038 artificial kidney) during the study period.
5. Having a record of dabigatran use for a purpose other than prevention of ischemic stroke and systemic embolism in non-valvular atrial fibrillation patients.
6. Having a record of dabigatran or warfarin before the hospitalization
7. Having a record of new diagnosis of atrial fibrillation after the initiation of dabigatran or warfarin treatment in the hospitalization period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japan
Sampling Method: Non-Probability Sample
Enrollment: 4313 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2016-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Japan (2):
  - 1160.254.81001 Boehringer Ingelheim Investigational Site, Shinagawa City
  - NISED Center, Tokyo, Shinagawa

RESULTS

PARTICIPANT FLOW:
Groups:
- Dabigatran Etexilate [Prazaxa®]: The patients were administered Dabigatran Etexilate 75 mg*2 mg capsules twice daily or 110 mg capsules twice daily orally for Non-Valvular Atrial Fibrillation (NVAF).
- Warfarin: Dose-adjusted Warfarin for several days to reach an effective International Normalized Ratio (INR) for ischemic stroke prevention due to NVAF.
Period: Overall Study
Arm/Group | Dabigatran Etexilate [Prazaxa®] | Warfarin
Started | 899 | 3414
Completed | 899 | 3414
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis set included patients who received the treatment Dabigatran Etexilate [Prazaxa®] or Warfarin.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate [Prazaxa®] | Warfarin | Total
Number analyzed (Participants) | 899 | 3414 | 4313
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (11.6) | 76.1 (10.4) | 74.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 297 | 1398 | 1695
  Male | 602 | 2016 | 2618

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay (LoS) From Treatment of Oral Anticoagulant Initiation to Hospital Discharge Without Consideration of Baseline
Description: The outcome measure presents LoS from initiation of treatment with oral anticoagulants to hospital discharge without consideration of baseline of patients hospitalized for any reason, who were subsequently treated with Dabigatran or Warfarin for a NVAF.
Time Frame: From the date of index treatment until the date of discharge from hospital, assessed upto 60 months.
Population: The analysis set included patients who received the treatment Dabigatran Etexilate [Prazaxa®] or Warfarin.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Dabigatran Etexilate [Prazaxa®] | Warfarin
Number analyzed (Participants) | 899 | 3414
Months | 9.8 (13.5) | 14.9 (19.4)
Statistical Analysis 1: Comparison: Dabigatran Etexilate [Prazaxa®] vs Warfarin; Test type: Superiority or Other; p < 0.001, Abadie-Imbens; LoS Average Treatment Effect on the Treated (ATET) [Dabigatran group], dispersion analysed with Abadie-Imbens's standard error; Mean = -2.484, 95% CI 2-sided [-3.717 to -1.251], Standard Error of Mean 0.629 — The ATET of LoS from oral anticoagulant initiation to hospital discharge was calculated as [Dabigatran - Warfarin] in the matched cohort of matching ratio 1:3

ADVERSE EVENTS:
Time Frame: Serious and other (non-serious) adverse events were not of interest in this study and therefore were not collected or assessed as part of the study, in addition individual patient data is not available therefore adverse event data is not presented.
Arm/Group | Dabigatran Etexilate [Prazaxa®] | Warfarin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No